CLINICAL TRIAL: NCT00461799
Title: Orlistat Treatment of Unconjugated Hyperbilirubinemia in Crigler-Najjar Disease; A Randomized Controlled Trial
Brief Title: Orlistat Treatment of Crigler-Najjar Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Erasmus Medical Center (Other); De Najjar Stichting (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CN-01
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Last update posted 2007-04-18 (Estimated); Status verified 2007-04

CONDITIONS: Crigler-Najjar Syndrome
Keywords: Crigler-Najjar disease.; Bilirubin.; Phototherapy.; Orlistat.; Unconjugated hyperbilirubinemia.
MeSH Terms: conditions — Crigler-Najjar Syndrome | interventions — Orlistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: orlistat

SUMMARY:
The purpose of this study was to determine whether orlistat is effective in decreasing plasma unconjugated bilirubin levels in patients with Crigler-Najjar disease.

DETAILED DESCRIPTION:
Unconjugated hyperbilirubinemia in Crigler-Najjar (CN) disease is conventionally treated with phototherapy and/or phenobarbital. Life-long daily phototherapy has considerable disadvantages. Main problems are a decreasing efficacy with age and a profound impact of the intensive phototherapy regimen on the quality of (social) life. An alternative treatment option for unconjugated hyperbilirubinemia is based on intestinal capture of UCB by oral treatment. Particularly when plasma UCB concentrations are high as in CN disease, UCB can diffuse from the blood into the intestinal lumen across the mucosa. Intestinal capture of UCB followed by fecal excretion reduces the enterohepatic circulation of UCB and subsequently decreases plasma UCB concentration. We demonstrated in Gunn rats, the animal model for CN disease, that orlistat treatment decreases plasma UCB concentrations parallel with increased fecal fat excretion, and induces net transmucosal excretion of UCB from the blood into the intestinal lumen. In human adults, orlistat has been widely applied for treatment of obesity, without serious side effects. Recent studies in obese adolescents and prepubertal children indicate that short-term orlistat treatment is well-tolerated by children and generally has only mild side effects. In the present randomized, placebo-controlled trial we determined in patients with CN disease the effects of orlistat treatment on plasma UCB concentrations, and on fecal excretion of fat and UCB.

ELIGIBILITY:
Inclusion Criteria:

* patients with Crigler-Najjar disease above the age of 7 years

Exclusion Criteria:

* cholestasis, chronic malabsorption syndrome, pregnancy

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16
Dates: Start 2003-09; Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
decrease in plasma unconjugated bilirubin level during orlistat
increase in fecal fat excretion during orlistat
increase in fecal bilirubin concentration during orlistat

CONTACTS AND LOCATIONS:
Overall Officials: Anja M. Hafkamp, MD, Principal Investigator — University Medical Center Groningen and Erasmus University Medical Center; Maarten Sinaasappel, MD, Study Chair — Erasmus Medical Center; Henkjan J. Verkade, MD, PhD, Study Director — University Medical Center Groningen
Locations (1):
- Erasmus University Medical Center, Rotterdam, Netherlands

REFERENCES:
- [Background] Hafkamp AM, Havinga R, Sinaasappel M, Verkade HJ. Effective oral treatment of unconjugated hyperbilirubinemia in Gunn rats. Hepatology. 2005 Mar;41(3):526-34. doi: 10.1002/hep.20589. PMID 15726662
- [Background] Hafkamp AM, Havinga R, Ostrow JD, Tiribelli C, Pascolo L, Sinaasappel M, Verkade HJ. Novel kinetic insights into treatment of unconjugated hyperbilirubinemia: phototherapy and orlistat treatment in Gunn rats. Pediatr Res. 2006 Apr;59(4 Pt 1):506-12. doi: 10.1203/01.pdr.0000203180.79636.98. PMID 16549520
- [Background] Nishioka T, Hafkamp AM, Havinga R, vn Lierop PP, Velvis H, Verkade HJ. Orlistat treatment increases fecal bilirubin excretion and decreases plasma bilirubin concentrations in hyperbilirubinemic Gunn rats. J Pediatr. 2003 Sep;143(3):327-34. doi: 10.1067/s0022-3476(03)00298-1. PMID 14517515
- [Background] Verkade HJ. A novel hypothesis on the pathophysiology of neonatal jaundice. J Pediatr. 2002 Oct;141(4):594-5. No abstract available. PMID 12378205